CLINICAL TRIAL: NCT00659399
Title: 07-742 Phase I/ Feasibility Study of Short Term Fondaparinux (Arixtra) in Chemotherapy-Pretreated Ovarian Carcinoma Patients at High Risk of Progression
Brief Title: Feasibility Study of Short Term Fondaparinux (Arixtra) in Chemotherapy-Pretreated Ovarian Carcinoma Patients at High Risk of Progression
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: NYU Langone Health (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Boris Kobrinsky, New York University Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-742
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Ovarian Carcinoma
Keywords: Pretreated Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fondaparinux — Arixtra 2.5 mg by subcutaneous injection once daily for 8 weeks or until disease recurrence or grade 3, 4 adverse events.
  Other Names: Arixtra; fondaparinux sodium

SUMMARY:
The purpose of this study is to assess feasibility and safety of using once daily Fondaparinux Sodium (ARIXTRA®) in patients with ovarian cancer who are in 'clinical remission' (no clinical evidence of disease) after chemotherapy but at high risk of ovarian cancer recurrence.

DETAILED DESCRIPTION:
Rationale:

A large body of work supports the association of abnormal coagulation (blood clot formation) and malignancy. A coagulation enzyme thrombin is able to 1) enhance cancer cell adhesion to platelets and endothelial cells 2) stimulate tumor cell growth, 3) increase metastasis and 4) stimulate tumor angiogenesis.

Thrombin inhibition has anti-metastatic and anti-tumor activity in mouse models. Recent meta-analysis of 4 major randomized clinical trials that have evaluated the effect of anticoagulants on overall survival in cancer patients comparing low molecular weight heparin (LMWH) to placebo demonstrates a 13% risk reduction in mortality at 1 year and 10% risk reduction at 2 years, which is statistically significant and independent of the potential confounding effect of anticoagulation in the prevention of venous thromboembolic disease.

Fondaparinux sodium (ARIXTRA® ) is a highly effective newer anticoagulant that is a fully synthetic pentasaccharide. Arixtra binds to antithrombin III and subsequently inhibits Factor Xa and hence thrombin generation. Arixtra has an excellent safety profile in clinical trials of over 10,000 patients. When compared to LMWHs, ARIXTRA® has a potential pharmacokinetic advantage based on its longer half-life of 16-17 hours.

Hypothesis:

The hypothesis to be tested is whether the completion of 8 weeks of ARIXTRA® in patients with ovarian cancer who are in 'clinical remission' (no clinical evidence of disease) after chemotherapy but at high risk of ovarian cancer recurrence is feasible and safe and if the inhibition of thrombin generation by ARIXTRA® in ovarian cancer will result in decrease ovarian cancer recurrence.

A concise description of the methodology:

The trial will be a prospective open-label cohort feasibility study of giving 2 months of ARIXTRA® in patients at high risk of recurrence of ovarian cancer. The planned accrual is 15 patients. Patients will be treated with a fixed dose of ARIXTRA® 2.5 mg by subcutaneous injection once daily. Treatment will continue for 2 months or until disease recurrence or grade 3 adverse events or patient refusal.

In addition, all patients will be followed for survival and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and ≤75 years of age
* Biopsy-proven ovarian, tubal or primary peritoneal epithelial adenocarcinomas;
* Performance status 0,1 (ECOG) ( table 2)
* Patients at high risk of clinical relapse: first remission stage III/IV who were suboptimally debulked (residual disease >1 cm)
* Patients of any stage who have recurred and are in second chemotherapy induced remission. Clinical remission defined as:

  * absence of symptoms that may be related to disease
  * imaging without abnormalities greater then or equal to 1 cm suspicious for disease (no ascites)
  * CA 125 obtained x 1 and <35 units/ml.
* Adequate end organ function, defined as the following:

  * Total bilirubin < 1.5 x ULN
  * SGOT and SGPT < 2.5 x UNL
  * Creatinine < 1.5 x ULN
  * ANC > 1.5 x 109/L
  * Platelets > 100 x 109/L
  * Weight ≥ 50 kg

Exclusion Criteria:

* Patients with performance status ECOG =2,3,4
* Patients who are on warfarin or prior therapeutic anticoagulation
* Patient has another primary malignancy that has required active intervention within 5 years, with the exception of basal cell skin cancer or a cervical carcinoma in situ.
* Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
* Patient who had a major surgery within 2 weeks prior to study entry
* Patients with the following lab abnormalities:

  * WBC <3000
  * absolute neutrophil count < 1,500
  * hemoglobin <10 g/dL
  * platelet < 100,000
  * creatinine clearance <30 cc/min
  * serum ALT, AST, or total bilirubin >1.5X the upper limit of normal
* Patients with known bleeding disorder

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Estimate the proportion of patients who complete an eight week course of once daily administration of fondaparinux (Arixtra). | 15 months

SECONDARY OUTCOMES:
Time to Recurrence | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Boris Kobrinsky, M.D., Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Cancer Institute Clinical Cancer Center, New York, New York, United States